CLINICAL TRIAL: NCT07120997
Title: A Prevention Strategy for the Indication of Prune Consumption in Perimenopausal Females: Can Prunes Attenuate Bone Loss?
Brief Title: Prunes Preventing Bone Loss in Perimenopause
Acronym: Prune-UP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: University of Georgia (Other); California Dried Plum Board (Other); United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mary Jane DeSouza, Distinguished Professor of Kinesiology and Physiology, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00027323; 14223973 (Other Grant/Funding Number: United States Department of Agriculture)
Record Dates: First submitted 2025-07-31; First posted 2025-08-13 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Perimenopausal Bone Loss
Keywords: Female; Transmenopause; Perimenopause; Perimenopausal Bone Loss; Menopause; Human; Osteoporosis; Non-pharmacologic therapy; Prune intake; Dried Plum
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcium and Vitamin D - Control group (Experimental): Participants will take calcium and vitamin D supplements daily for a baseline period and for the duration of the intervention. Participants will be asked to refrain from consumption of prunes and fruits that have high phenolic content for the duration of the intervention (18 months).
  Interventions: Dietary Supplement: Calcium supplement; Dietary Supplement: Vitamin D Supplement
- 50g Prunes, Calcium, and Vitamin D - Intervention Group (Experimental): Participants will take calcium and vitamin D supplements daily for a baseline period and for the duration of the intervention. Additionally, participants will be provided with prunes and asked to consume 6 (50g) prunes per day for the duration of the intervention (18 months).
  Interventions: Dietary Supplement: Prunes; Dietary Supplement: Calcium supplement; Dietary Supplement: Vitamin D Supplement

INTERVENTIONS:
Dietary Supplement: Prunes — Participants randomized to the 50g prune group will consume 6 prunes per day for the duration of the 18-month intervention.
  Arms: 50g Prunes, Calcium, and Vitamin D - Intervention Group
Dietary Supplement: Calcium supplement — All participants will consume calcium supplements daily for a baseline period and for the duration of the 18-month intervention.
Dietary Supplement: Vitamin D Supplement — All participants will consume Vitamin D supplements daily for a baseline period and for the duration of the 18-month intervention.

SUMMARY:
Dietary interventions of prune consumption during the transmenopausal period are innovative methods to prevent bone loss. Modern medicine does not intervene to prevent or attenuate this highly vulnerable period of bone loss which, if successfully attenuated, can potentially prevent/delay osteoporosis in women. The transmenopausal period represents an opportunistic window for the study because bone loss is at its greatest at this time, with females losing as much as 6-7% of bone. If this project is successful at attenuating bone loss, it can immediately be disseminated to the public to promote prune consumption to slow down and attenuate perimenopausal bone loss. As such, this project could improve the long-term bone health of females and avoid or delay osteoporosis and improve quality of life. The long-term goal of this study is to test the novel hypothesis that prune consumption for 18 months during the 3-year transmenopausal period prevents the dramatic rate of bone loss in perimenopausal females during a window of heightened physiological vulnerability. At Penn State University, the study will compare the effects of 18 months of daily dietary consumption of 50 g of prunes (5-6) versus a no-prune control group on bone outcomes (bone mineral density, bone geometry), mechanistic factors (bone and inflammatory markers, inflammatory response of ex vivo cultured peripheral blood mononuclear cells, monocytes), and gut microbiome.

DETAILED DESCRIPTION:
Females spend at least one-third of their lifespan after menopause, therefore strategies that improve the long-term health of women and engage a prevention strategy to improve health are warranted and represent opportunities for high impact and high return on investment. After menopause, one in two females will suffer a fragility fracture in their lifetime, and the mortality rate after a hip fracture is as high as 25%. Moreover, since osteoporosis-related treatment costs more than $100 billion worldwide, strategies that focus on the prevention of osteoporosis-related fragility fractures are warranted. As such, the prevention of bone loss, osteoporosis, and its related fractures is much preferred over treatment of osteoporosis given the high costs, negative side effects, and poor compliance to pharmacological treatment regimens. Therefore, research addressing the optimization of the health of perimenopausal females to delay chronic disease is very much necessary and represents the overall objective of this project. Given the high mortality rate of hip fractures, this intervention may potentially save people's lives while reducing a significant healthcare burden.

The long-term goal of this project is to change the course of bone loss during a very specific and opportunistic intervention window, i.e., the transmenopausal window. This window of intervention is opportunistic because females lose more bone at the hip and spine than at any other time; that is, as much as 6% and 7% at the hip and spine, respectively. In fact, the amount of bone loss during this three-year transmenopausal window that initiates late perimenopause is greater than the amount of bone loss observed during the postmenopause window, when the latter is defined as 2 to 5 years after the final menstrual period. The STRAW+10 investigators defined the stages of menopause, including the transmenopause period, a stage in life that is associated with dramatic bone loss. As such, this project is novel, innovative, and can potentially delay the serious effects of osteoporotic bone loss and associated fractures, to which transmenopausal bone loss significantly contributes. When one considers that as of 2021, there were approximately 1.02 billion females over 50 years of age worldwide, with an estimated 1.2 billion females over the age of 50 by 2030, accounting for 26% of all females worldwide, the potential impact of this project is substantial. Indeed, this project may affect the long-term picture of bone health for millions of females by delaying or attenuating the acceleration of bone loss during the transmenopause period. Moreover, since osteoporosis affects millions of females worldwide, this project has the potential to offset the devasting long-term effects of accelerated bone loss during transmenopause that is associated with osteoporosis.

The overall objective of this research is to test whether prunes are effective in attenuating the rapid transmenopausal bone loss observed in late peri and early postmenopausal females. The investigators will study the effects of 18 months of prune consumption in females recruited during the late peri and early postmenopausal stage, allowing a high probability for data collection spanning the transmenopausal period of heightened bone loss, i.e., 12 months before the final menstrual period and the two years following the final menstrual period. The investigators will also examine the physiological mechanisms underlying the bone trophic effects of prune consumption to seek evidence on how prunes work. If successful, prunes will be demonstrated to be a powerful strategy to attenuate and delay the rapid decline in bone mineral density and decrements in microarchitecture that eventually lead to osteoporosis and heightened risk for fracture.

ELIGIBILITY:
Inclusion Criteria:

* Age 44 to 55 years
* Not severely obese (BMI <35 kg/m^2)
* Healthy (determined by a screening questionnaire, physical and medical history by a certified nurse practitioner, complete metabolic panel, and complete blood count)
* Willing to include prunes in their daily diet
* Not taking any natural dietary supplement containing phenolics, i.e.,< 1 cup/day of blueberries or apples for at least 2 months prior to study entry
* Non-smoking
* Ambulatory
* No menses for ≥60 days but not more than 18 months post final menstrual period
* Only participants who have a determinable natural (not surgical) final menstrual period date are eligible

Exclusion Criteria:

* Subjects who regularly consume prunes, dried apples, prune juice, or heavy consumers of blueberries (1 cup or more/day)
* History of vertebral fracture or fragility fracture of the wrist, humerus, hip or pelvis after age 45 yr)
* Untreated hyper- or hypothyroidism
* Current hyper- or hypoparathyroidism
* Significantly impaired renal function
* Current hypo- or hypercalcemia
* History of spinal stenosis
* History of heart attack, stroke, thromboembolism, kidney disease, malabsorption syndrome, or seizure disorders
* Positive for HIV, Hep-C or Hep-B surface antigen and malignancy
* Use of the following agents affecting bone metabolism: intravenous bisphosphonates at any time; fluoride (for osteoporosis) within the past 24 months; denosumab at any time; bisphosphonates, parathyroid hormone or strontium within the past 12 months; calcitonin; selective estrogen receptor modulators within the past 12 months; systemic oral or transdermal estrogen within the past 3 months; systemic glucocorticosteroids (≥ 5 mg prednisone equivalent per day for more than 10 days); or tibolone within the past 3 months
* Hormonal contraception within the past three months
* Subjects who will not consume study provided dietary items or who will not stop taking their own natural product supplements

Ages: 44 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in areal bone mineral density (via DXA) of the lumbar spine, total hip, and femoral neck | Baseline, month 9, month 18
  Percent change in areal bone mineral density measured at baseline, month 9, and month 18 of the 18-week dietary intervention at the lumbar spine, total hip, and femoral neck.

SECONDARY OUTCOMES:
Changes from baseline in Spine Trabecular Bone Score (TBS) (via DXA) | Baseline, month 9, and month 18
  Changes in Spine Trabecular Bone Score (TBS) assessed at baseline, month 9, and month 18 of the 18-month dietary intervention from lumbar spine DXA scans. The measurements will provide additional information about the effects of the intervention on trabecular bone.
Percent change from baseline in volumetric BMD of the tibia and radius (via pQCT) | Baseline, month 9, and month 18
  Percent change in volumetric BMD, cortical and trabecular compartments, measured during baseline, month 9, and month 18 of the 18-month dietary intervention at the tibia and radius. The combination of measurements will provide an overall picture of the 3-dimensional structure of a weight bearing (tibia) and non-weight bearing (radius) site and how the sites are impacted by the intervention.
Percent change from baseline in bone geometry measurements of the tibia and radius (via pQCT) | Baseline, month 9, and month 18
  Percent change in bone geometry estimates (total bone area, cortical and trabecular area, cortical thickness) measured during baseline, and month 9, and month 18 of the 18-month dietary intervention at the tibia and radius. The combination of measurements will provide an overall picture of the 3-dimensional structure of a weight bearing (tibia) and non-weight bearing (radius) site and how the sites are impacted by the intervention.
Percent change from baseline in bone strength index of the tibia and radius (via pQCT) | Baseline, month 9, and month 18
  Percent change in bone strength index (BSI) measured during baseline, and month 9, and month 18 of the 18-month dietary intervention at the tibia and radius. The measurement will provide an overall picture of bone strength and of the 3-dimensional structure of a weight bearing (tibia) and non-weight bearing (radius) site and how the sites are impacted by the intervention.
Percent change from baseline in stress strain index of the tibia and radius (via pQCT) | Baseline, Month 9, Month 18
  Percent change in stress strain index (SSI), a bone strength measurement, measured during baseline, month 9, and month 18 of the 18-month dietary intervention at the tibia and radius. The measurements will provide an overall estimate of bone strength of a weight bearing (tibia) and non-weight bearing (radius) site and how the sites are impacted by the intervention.
Percent change from baseline in polar moment of inertia measurements of the tibia and radius (via pQCT) | Baseline, Month 9, Month 18
  Percent change in polar moment of inertia (section modulus) measured during baseline, and month 9, and month 18 of the 18-month dietary intervention at the tibia and radius. The measurement will provide an overall picture of the 3-dimensional structure and bone strength of a weight bearing (tibia) and non-weight bearing (radius) site and how the sites are impacted by the intervention.
Change from baseline in C-terminal telopeptide of type I collagen (CTx) | Baseline, month 9, and month 18
  Change in serially-sampled fasting serum concentrations of C-terminal telopeptide of type I collagen (CTx), a marker of bone resorption, at baseline, month 9, and month 18 of the 18-month dietary intervention. Changes in bone resorption markers will assist in understanding the underlying mechanisms behind changes in the rates of bone resorption.
Change from baseline in Tartrate-resistant acid phosphatase (Trap 5b) | Baseline, month 9, and month 18
  Change in serially-sampled fasting serum concentrations of Tartrate-resistant acid phosphatase (Trap 5b), a marker of bone resorption, at baseline, month 9, and month 18 of the 18-month dietary intervention. Changes in bone resorption markers will assist in understanding the underlying mechanisms behind changes in the rates of bone resorption.
Change from baseline in expression of inflammatory markers | Baseline, month 9, and month 18
  Change in lipopolysaccharide(LPS)-stimulated peripheral blood mononuclear cell (PBMC) gene expression of inflammatory markers (interleukin-1β, interleukin-6, and tumor necrosis factor-α) at baseline, month 9, and month 18 of the dietary intervention. Additionally, the relationship between the changes in gene expression of inflammation markers and bone outcomes will be explored. The combined changes of the gene expression of inflammatory markers will provide a comprehensive picture of the inflammatory environment of the participants before, during and following the dietary intervention. This comprehensive picture will assist in understanding the mechanisms by which the inflammatory environment contributes to bone loss in transmenopause and how the dietary intervention impacts those factors.
Change from baseline in gut permeability | Baseline, month 9, and month 18
  Change in serially-sampled fasting serum concentrations of zonulin, a gut permeability marker, at baseline, month 9, and month 18 of the 18-month dietary intervention. Changes in zonulin will assist in understanding the underlying mechanisms of changes in the gut and bone metabolism.
Change from baseline in gut microbiome | Baseline, month 9, and month 18
  Serially-sampled stool samples for assessment of changes in the Beta diversity of gut microbiome at baseline, month 9, and month 18 of the 18-month dietary intervention. Additionally, the relationship between the changes in the gut microbiome and bone outcomes will be explored.

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Health and Exercise Laboratory, The Pennsylvania State University, University Park, Pennsylvania, United States